CLINICAL TRIAL: NCT01104675
Title: A Phase 2 Study of Oral ENMD-2076 Administered to Patients With Platinum Resistant Ovarian Cancer
Brief Title: Study of Oral ENMD-2076 Administered to Patients With Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2076-CL-004
Record Dates: First submitted 2010-04-14; First posted 2010-04-15 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Ovarian Cancer; Fallopian Cancer; Peritoneal Cancer
Keywords: ovarian; platinum resistant ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — ENMD 2076

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ENMD-2076 treatment (Experimental)
  Interventions: Drug: ENMD-2076

INTERVENTIONS:
Drug: ENMD-2076 — 275 mg (or 250 mg for BSA < 1.65) per day in oral capsules in 28 day continuous cycles

SUMMARY:
The purpose of this study is to determine whether oral ENMD-2076 is effective in treatment of patients with platinum resistant ovarian, fallopian, or peritoneal cancer. Additional sites to be added.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically documented diagnosis of ovarian, fallopian or peritoneal cancer that is platinum resistant.
* Have a pre-study echocardiogram or multigated acquisition (MUGA) scan with an actual left ventricular ejection fraction of greater than or equal to the institution lower limit of normal
* Greater than or equal to 18 years of age
* Have clinically acceptable laboratory screening results
* Have an ECOG performance status of 0 or 1
* Able to tolerate oral medications

Exclusion Criteria:

* Have uncontrolled hypertension (systolic blood pressure greater than 150mmHg or diastolic blood pressure greater than 100mmHg); require two or more antihypertensive medications to control hypertension (including ACE inhibitors, beta blockers, calcium channel blockers, or diuretics)
* Have chronic atrial fibrillation or QTc interval corrected for heart rate of greater than 470 msec
* Have active, acute, or chronic clinically significant infections or bleeding
* Have persistent 2+ protein by urinalysis or a history of nephrotic syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William Gannon, MD, MBA, Study Director — CASI Pharmaceuticals, Inc.
Locations (6):
- United States (5):
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Dana Farber/Partners Cancer Care, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
- Princess Margaret Hospital, Toronto, Ontario, Canada